CLINICAL TRIAL: NCT06732505
Title: A Phase I Study to Assess the Safety and Efficacy of [225Ac]Ac-DOTATATE in Patients With Inoperable, Locally Advanced or Metastatic, Progressive, Well-Differentiated,SSTR+ GEP-Nens
Brief Title: A Phase I Study to Assess the Safety and Efficacy of [225Ac]Ac-DOTATATE in Patients With SSTR+ GEP-Nens
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Sinotau Pharmaceutical Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IIT-XT024-1-01
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Neuroendocrine Neoplasm
Keywords: [225Ac]Ac-DOTATATE; neuroendocrine neoplasm
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [225Ac]Ac-DOTATATE (Experimental): Investigational radiotherapeutic drug targeting somatostatin receptor-positive neuroendocrine neoplasms in PRRT naive patients (Cohort 1) and previous PRRT patients (Cohort 2)
  Interventions: Drug: [225Ac]Ac-DOTATATE

INTERVENTIONS:
Drug: [225Ac]Ac-DOTATATE — The dose escalation phase will be divided into two cohorts: patients who had previously received 177Lu-PRRT will be enrolled in cohort 1, and patients who had not received 177Lu-PRRT will be enrolled in cohort 2. Dose escalation was performed independently in the two cohorts. DL1 will be administered as a dose of 90kBq/kg per cycle, and DL2 will be administered as a single dose of 120kBq/kg per cycle.Every patient will receive one [225Ac]Ac-DOTATATE infusion every 8 weeks for up to 4 cycles.
  The dose expansion phase will be divided into 3 cohorts based on Ki-67 index.

SUMMARY:
This is a phase I study to assess the safety and efficacy of [225Ac]Ac-DOTATATE in patients with inoperable, locally advanced or metastatic, progressive, Well-Differentiatedwell differentiated, somatostatin receptor positive gastroenteropancreatic neuroendocrine neoplasms with either no prior history of peptide receptor radionuclide therapy (PRRT naive) or prior history of peptide receptor radionuclide therapy (Previous PRRT).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have the ability to understand and sign an approved informed consent form (ICF).
2. Patients must be >= 18 and <＝80 years of age.
3. Histopathologically confirmed G1 or G2 or G3 GEP-NET or GEP-NEC；
4. Unresectable locally advanced or metastatic GEP-NET which confirmed by imaging examination.
5. G1 or G2 NET patients: previously received fixed-dose Octreotide LAR (20-30 mg/3-4 weeks) for at least 12 weeks of continuous treatment with disease progression;G3 NET orNEC patients: previously received at least 1 line therapy with disease progression.
6. Presence of at least 1 measurable site of disease (based on RECIST 1.1).
7. SSTR-PET positive.
8. ECOG score of 0 or 1.
9. Life expectancy of at least 12 weeks.
10. Sufficient bone marrow capacity and organ function:

    Serum creatinine ≤1.5×ULN or creatinine clearance ≥50 ml/min (Cockcroft Gault formula).

    Hemoglobin≥90g/L, neutrophil count ≥1.5×10^9/L, platelets≥100×10^9/L. Serum total bilirubin ≤1.5×ULN. Serum albumin ≥30g/L. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 2.5×ULN，or ALT/AST≤5×ULN with liver metastases.

    Partially activated prothrombin time (APTT) ≤1.5 x ULN.
11. Subjects of childbearing potential voluntarily use an effective method of contraception, such as condoms, oral or injectable contraceptives, IUDs, etc., during treatment and within 6 months of the last use of the trial drug.

Exclusion Criteria:

1. Pregnant or lactating females.
2. Received the following treatments within 4 weeks prior to initiation of study treatment, including but not limited to surgery (except biopsy), radical radiotherapy, hepatic artery interventional embolization, cryoablation of liver metastases, or radiofrequency ablation.
3. Received systemic antitumor therapy such as targeted therapy, immunotherapy, antitumor herbal therapy, chemotherapy within 4 weeks prior to initiation of study treatment.
4. Rapid progression with previous PRRT therapy.
5. Any patient receiving treatment with short-acting Octreotide, which cannot be interrupted for 24 h before and 24 h after the administration of initiation of study treatment, or any patient receiving treatment with Octreotide LAR, which cannot be interrupted for at least 6 weeks before the administration of initiation of study treatment.
6. Toxicity of prior antitumor therapy has not returned to ≤ grade 1 levels (except for alopecia).
7. Received external beam radiation therapy for bone metastases within 2 weeks prior to initiation of study treatment.
8. Known brain metastases, unless these metastases have been treated and stabilized for at least 24 weeks, prior to enrollment in the study.
9. Uncontrolled congestive heart failure.
10. uncontrolled diabetes mellitus, including baseline fasting glucose > 2 x ULN.
11. Known other malignancies (except for those without recurrence within 5 years after adequate treatment).
12. Known hypersensitivity to Lutetium[177Lu] Oxodotreotide Injection or [225Ac]Ac-DOTATATE Injection and their excipients.
13. Known to be unsuitable for enhanced CT or MRI contrast imaging due to allergic reaction or renal insufficiency.
14. Any clinically significant active infection.
15. Participated in other drug clinical trials within 4 weeks prior to initiation of study treatment and received treatment with the corresponding trial drug.
16. Any other disease, mental status or surgical condition that is uncontrolled, may interfere with study completion (including poor compliance) or is inappropriate for the use of the investigational drug.
17. Other treatment options (e.g., chemotherapy, targeted therapy) that, in the opinion of the investigator, are more appropriate for the patient than the treatment provided in the study based on the patient's disease characteristics.
18. Unsuitable for the study for any reason, in the opinion of the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-09-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of 225Ac-DOTATATE | 32 weeks following first 225Ac-DOTATATE injection
  Incidence and severity of adverse events (AEs) according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0
Recommended phase II dose of 225Ac-DOTATATE | First 56 days following first 225Ac-DOTATATE injection
  Rate incidence of dose-limiting toxicities (DLT)

SECONDARY OUTCOMES:
ORR | 24 months after last dose administration
  ORR was calculated as the proportion of patients with tumour size reduction (sum of partial responses (PR) and complete responses (CR)) and assessed by investigator according to RECIST 1.1.
PFS | 24 months after last dose administration
  PFS will be defined as the number of days from the first dose of [225Ac]-DOTATATE to documented tumor progression per RECIST 1.1 criteria or death due to any cause.
DoR | 24 months after last dose administration
  DoR was defined as the time from initially meeting the criteria for response (CR or PR) until the time of progression and assessed by investigator according to RECIST 1.1.
TTP | 24 months after last dose administration
  TTP was defined as the time from randomization to progression assessed by investigator. It included patients who dropped out due to toxicity, but omitted patients who died without measured progression (censored to last follow-up date or death date).
DCR | 24 months after last dose administration
  DCR is defined as the incidence of complete response, partial response and stable disease assessed by investigator according to RECIST v1.1.
12-month PFS Rate | From date of enrollment until date of progression or date of death from any cause, whichever comes first，assessed up to approximately 24 months
  12-month Progression-Free Survival rate was defined as the proportion of patients whose time from enrollment to disease progression according to RECIST v1.1 or death exceeds 12 months.

OTHER OUTCOMES:
Whole body and organ uptake of [225Ac]Ac-DOTATATE | 8 weeks after the first dose administration
  To estimate the absorbed doses of target organs and lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No